CLINICAL TRIAL: NCT02019719
Title: A 4-Week, Phase II, Randomized, Double-Blind, Dose-Ranging, Placebo-Controlled, Parallel-Group, Multi-Center Study to Evaluate the Safety, Efficacy and Pharmacokinetics of GSK1278863 in Japanese Hemodialysis-Dependent Subjects With Anemia Associated With Chronic Kidney Disease
Brief Title: Study to Evaluate the Safety, Efficacy and Pharmacokinetics of GSK1278863 in Japanese Hemodialysis-Dependent Subjects With Anemia Associated With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116099
Record Dates: First submitted 2013-10-31; First posted 2013-12-24 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Anaemia
Keywords: Hemodialysis; GSK1278863; Pharmacokinetics; Erythropoiesis Stimulating Agents; Chronic Kidney Disease; Hemoglobin; Recombinant Erythropoietin; Prolyl Hydroxylase Inhibitor; Anemia
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- GSK1278863 4 milligrams (mg) (Experimental): Subjects will receive GSK1278863 4 mg once daily for 4 weeks
  Interventions: Drug: GSK1278863
- GSK1278863 6 mg (Experimental): Subjects will receive GSK1278863 6 mg once daily for 4 weeks
  Interventions: Drug: GSK1278863
- GSK1278863 8 mg (Experimental): Subjects will receive GSK1278863 8 mg once daily for 4 weeks
  Interventions: Drug: GSK1278863
- GSK1278863 10 mg (Experimental): Subjects will receive GSK1278863 10 mg once daily for 4 weeks
  Interventions: Drug: GSK1278863
- Placebo (Placebo Comparator): Subjects will receive placebo once daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1278863 — GSK1278863 will be supplied as film coated tablets for oral administration containing 1 mg, 2 mg, or 5 mg of GSK1278863.
  Arms: GSK1278863 10 mg; GSK1278863 4 milligrams (mg); GSK1278863 6 mg; GSK1278863 8 mg
Drug: Placebo — Film coated tablets of GSK1278863 matching placebo for oral administration.
  Arms: Placebo

SUMMARY:
This study aims to characterize the relationship between dose of GSK1278863 and hemoglobin (Hgb) response in hemodialysis-dependent (HDD) subjects with anemia associated with chronic kidney disease (CKD). It is anticipated that the data generated will enable selection of the starting dose(s) and optimize dose adjustment regimen(s) for Phase 3 clinical trials. This study will consist of a screening phase of 3-9 weeks, a 4-week treatment phase and a follow-up visit approximately 4 weeks after completing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age (Informed concent): Japanese >=20 years of age
* Gender (Screening 2 verification only): Female and male
* Females: must be of childbearing potential, and must agree to use one of the approved contraception methods from Screening 2 until completion of the Follow-up Visit. OR Of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrea [in questionable cases a blood sample with simultaneous follicle stimulating hormone 23.0 - 116.3 million international units (MIU)/millilitre (mL) and estradiol <= 10 picograms (pg)/mL is confirmatory]. Females on hormone replacement therapy (HRT) whose menopausal status is in doubt will be required to use one of the approved contraception methods if they wish to continue their HRT during the study. Otherwise they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method. Males: must agree to use one of the approved contraceptive methods from the time of Screening 2 until completion of the Follow-up Visit.
* Corrected QT interval (QTc) (Screening 2 verification only): Bazett's Correction of QT Interval (QTcB) <470 milliseconds (msec) or QTcB <480 msec in subjects with bundle branch block. There is no QTc inclusion criterion for a subject with a predominantly paced rhythm.
* Dialysis frequency: On hemodialysis (HD) three times weekly for at least 8 weeks prior to Screening 2 through Day 1.
* Dialysis adequacy (Screening 2 only): A single-pool Kt/Vurea of 1.2 based on a historical value obtained within the prior month in order to ensure the adequacy of dialysis. If Kt/Vurea is not available, then an average of the last 2 values of urea reduction ratio (URR) of at least 65%.
* Hemoglobin: Target stable Hgb between 9.5-12.0 g/dL at screening.
* Stable erythropoiesis-stimulating agent (ESA) dose (Screening 2 only): Using the same ESA (epoetins or their biosimilar, or darbepoietin) with total weekly doses that varied by no more than 50% during the 4 weeks prior to Screening 2.
* Iron replacement therapy: Subjects may be on stable maintenance oral or intravenous (IV) (<100 milligrams [mg]/week) iron supplementation. If subjects are on oral or IV iron, then doses must be stable for the 4 weeks prior to Screening 2, and Screening 2 through Week 4.

Exclusion Criteria:

* Dialysis modality: Planned change from HD to peritoneal dialysis within the study time period.
* Renal transplant: Renal transplant anticipated or scheduled within the study time period.
* High ESA dose (Screening 2 verification only): As defined by an epoetin dose of >=360 IU/kilograms (kg)/week IV or darbepoetin dose of >=1.8 micrograms (μg)/kg/week IV within the prior 8 weeks through Screening 2.
* methoxy polyethylene glycol epoetin beta (Screening 2 verification only): Use of methoxy polyethylene glycol epoetin beta within the prior 8 weeks through Screening 2.
* Vitamin B12: At or below the lower limit of the reference range
* Folate: <2.0 nanograms (ng)/mL (<4.5 nanomoles [nmol]/liters [L])
* Iron status: Ferritine <100 ng/mL (<100 μg/L) AND Transferrin saturation (TSAT) <20%
* Myocardial infarction or acute coronary syndrome: Within the 8 weeks prior to Screening 2 through Day 1.
* Stroke or transient ischemic attack: Within the 8 weeks prior to Screening 2 through Day 1.
* Heart failure: Class III/IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system or symptomatic right heart failure diagnosed prior to Screening 2 through Day 1.
* Hypertension: Defined using pre-dialysis vitals of diastolic blood pressure >100 mmHg or systolic blood pressure >170 mmHg.
* Thrombotic disease: History of thrombotic disease (e.g., venous thrombosis such as deep vein thrombosis or pulmonary embolism, or arterial thrombosis such as new onset or worsening limb ischemia requiring intervention), except vascular access thrombosis, within the 8 weeks prior to Screening 2 through Day 1
* Eyes: History of proliferative retinopathy requiring treatment within the prior 12 months or macular edema requiring treatment..
* Inflammatory disease: Active chronic inflammatory disease that could impact erythropoiesis (e.g., scleroderma, systemic lupus erythematosis, rheumatoid arthritis, celiac disease) diagnosed prior to Screening 2 through Day 1.
* Hematological disease: Any hematological disease including those affecting platelets, white or red blood cells (e.g. sickle cell anemia, myelodysplastic syndromes, hematological malignancy, myeloma, hemolytic anemia and thalassemia), coagulation disorders (e.g., antiphospholipid syndrome, Protein C or S deficiency), or any other cause of anemia other than renal disease diagnosed prior to Screening 2 through Day 1.
* Liver disease: Current liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or evidence at Screening of abnormal liver function tests [alanine transaminase (ALT) or aspartate transaminase (AST) >2.0 x upper limit of normal (ULN) or total bilirubin > 1.5 x ULN]; or other hepatic abnormalities that in the opinion of the investigator (subinvestigator) would preclude the subject from participation in the study.
* Major surgery: Major surgery (excluding vascular access surgery) within the prior 8 weeks, within the Screening 2 to Day 1 or planned during the study.
* Transfusion: Blood transfusion within the prior 8 weeks, within the Screening 2 to Day 1 or an anticipated need for blood transfusion during the study.
* Gastrointestinal (GI) bleeding: Evidence of actively bleeding peptic, duodenal, or esophageal ulcer disease OR clinically significant GI bleeding within the 8 weeks prior to Screening 2 through Day 1.
* Acute infection: Clinical evidence of acute infection or history of infection requiring IV antibiotic therapy within 8 weeks prior to Screening 2 through Day 1.
* Malignancy: Subjects with a history of malignancy within the prior 5 years, who receiving treatment for cancer, or who have a strong family history of cancer (e.g., familial cancer disorders); with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated prior to Screening 2 through Day 1.
* Severe allergic reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product
* Drugs and supplements: Use of any prescription or non-prescription drugs or dietary supplements that are prohibited from Screening 2 until the Follow-up Visit.
* Prior investigational product exposure: The Subject has participated in a clinical trial and has received an experimental investigational product within the prior 30 days from Screening 2 through Day 1.
* Pregnancy or lactation: Pregnant females as determined by positive serum Human Chorionic Gonadotrophin (hCG) test (Screening 2 only) OR women who are lactating at Screening 2 and/or Day 1 or during the trial.
* Other conditions: Any other condition, clinical or laboratory abnormality, or examination finding that the Investigator would consider inappropriate to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2014-08-06 (Actual); Study Completion 2014-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Japan (12):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Toyama

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 116099 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116099 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116099 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116099 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116099 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116099 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116099 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a study to evaluate dose-response of GSK1278863 in approximately 95 Japanese Hemodialysis-dependent (HDD) participants with anemia associated with Chronic Kidney Disease (CKD) conducted across 21 centers in Japan from 05 November 2013 to 06 August 2014.
Pre-assignment Details: This study consisted of a screening phase of 3-9 Week , a 4 Week treatment phase and a follow-up visit that occurred approximately 4 Week after completing treatment. Study completion was defined as completing the final visit including those in the follow-up period.
Groups:
- Placebo: Eligible participant's received matching placebo to GSK1278863 once daily for the 4 Week treatment period.
- GSK1278863 4 mg: Eligible participant's received GSK1278863 4 milligrams (mg) once daily for the 4 Week treatment period.
- GSK1278863 6 mg: Eligible participant's received GSK1278863 6 mg once daily for the 4 Week treatment period.
- GSK1278863 8 mg: Eligible participant's received GSK1278863 8 mg once daily for the 4 Week treatment period.
- GSK1278863 10 mg: Eligible participant's received GSK1278863 10 mg once daily for the 4 Week treatment period.
Period: Overall Study
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Started | 19 | 19 | 20 | 19 | 20
Completed | 13 | 18 | 20 | 17 | 18
Not Completed | 6 | 1 | 0 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0
Not completed — Protocol defined stopping criteria | 2 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK1278863 4 mg: Eligible participant's received GSK1278863 4 mg once daily for the 4 Week treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | Total
Number analyzed (Participants) | 19 | 19 | 20 | 19 | 20 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (8.98) | 61.6 (8.49) | 58.9 (9.90) | 66.0 (9.23) | 62.2 (11.13) | 62.4 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 8 | 12 | 9 | 47
  Male | 12 | 8 | 12 | 7 | 11 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 19 | 19 | 20 | 19 | 20 | 97
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (CFB) in Hemaglobin (Hgb) at Week 4
Description: Baseline was defined as the value on Day 1. CFB was calculated by subtracting the baseline value from the post-dose value at Week 4. To model the dose-response relationship a four-parameter Emax model was used. E0 is the expected Hgb change from Baseline for a participant receiving placebo and experiencing the average Hgb Baseline observed in the study. Emax is the expected Hgb change from Baseline for a participant receiving the highest dose above which no further increase in response can be achieved. ED50 is the dose that attains the intermediate response. Gamma is the slope parameter. Minimal Effective Dose (MED) is defined as the smallest dose that achieves a placebo-corrected change of 0.5 g/dL over Week 4. Target dose (TD) is defined as the dose that achieves a placebo-corrected 1.0 g/dL change over Week 4. Maximum Acceptable Dose (MAD) is defined as the dose that achieves a placebo-corrected 2.0 g/dL change over Week 4.
Time Frame: Baseline (Day 1) and Week 4
Population: Intent-to-Treat (ITT) population comprised of all randomized participants who received at least one dose of study drug, had a Baseline and at least one corresponding on treatment assessment. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: grams/deciliter (g/dL)
Groups:
- Placebo: Eligible participant's received matching placebo to GSK1278863 once daily for the 4W treatment period.
- GSK1278863 4 mg: Eligible participant's received GSK1278863 4 mg once daily for the 4 weeks treatment period.
- GSK1278863 6 mg: Eligible participant's received GSK1278863 6 mg once daily for the 4 weeks treatment period.
- GSK1278863 8 mg: Eligible participant's received GSK1278863 8 mg once daily for the 4 weeks treatment period.
- GSK1278863 10 mg: Eligible participant's received GSK1278863 10 mg once daily for the 4 weeks treatment period.
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 15 | 18 | 20 | 18 | 19
grams/deciliter (g/dL) | -1.52 (0.212) | -0.29 (0.200) | -0.02 (0.193) | 0.60 (0.202) | 0.92 (0.196)
Statistical Analysis 1: Comparison: Placebo vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg; Test type: Superiority or Other; E0 (g/dL) = -1.37, 95% CI 2-sided [-1.72 to -1.03] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 2: Comparison: Placebo vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg; Test type: Superiority or Other; ED50 (mg) = 21.88, 95% CI 2-sided [9.99 to 42.64] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 3: Comparison: Placebo vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg; Test type: Superiority or Other; Emax (g/dL) = 5.88, 95% CI 2-sided [3.20 to 8.61] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 4: Comparison: Placebo vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg; Test type: Superiority or Other; Gamma = 1.13, 95% CI 2-sided [0.70 to 1.68] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 5: Comparison: Placebo vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg; Test type: Superiority or Other; Var = 0.66, 95% CI 2-sided [0.50 to 0.88] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 6: Comparison: Placebo vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg; Test type: Superiority or Other; MED (mg) = 1.98, 95% CI 2-sided [0.75 to 3.41] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 7: Comparison: Placebo vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg; Test type: Superiority or Other; TD (mg) = 3.90, 95% CI 2-sided [2.20 to 5.63] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 8: Comparison: Placebo vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg; Test type: Superiority or Other; MAD (mg) = 8.65, 95% CI 2-sided [6.51 to 11.44] — Posterior median and 95% credibility intervals were estimated using Bayesian methods

2. Secondary Outcome: CFB in Hgb Upto Week 8
Description: Hgb assessments were performed at Baseline, Week 1, Week 2, Week 3, W eek4/Early withdrawal and Week 8 (follow-up) based on central laboratory (Quest diagnosis). Baseline was defined as the value on Day 1. CFB was calculated by subtracting the Baseline value from the post-dose value at Week 4.
Time Frame: Baseline (Day 1) Upto Week 8
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
g/dL
  CFB at Week 1: number analyzed (Participants) | 17 | 19 | 20 | 19 | 20
  CFB at Week 1 | -0.34 (0.485) | -0.23 (0.374) | -0.35 (0.462) | -0.31 (0.481) | -0.17 (0.318)
  CFB at Week 2: number analyzed (Participants) | 17 | 18 | 20 | 18 | 19
  CFB at Week 2 | -0.79 (0.538) | -0.32 (0.449) | -0.32 (0.780) | 0.01 (0.586) | 0.24 (0.353)
  CFB at Week 3: number analyzed (Participants) | 15 | 18 | 20 | 18 | 19
  CFB at Week 3 | -1.14 (0.743) | -0.42 (0.658) | -0.34 (0.776) | 0.21 (0.692) | 0.37 (0.471)
  CFB at Week 4: number analyzed (Participants) | 13 | 18 | 20 | 18 | 18
  CFB at Week 4 | -1.31 (0.923) | -0.33 (0.754) | -0.22 (1.008) | 0.34 (1.069) | 0.51 (0.679)
  CFB at Week 8, Follow-up: number analyzed (Participants) | 5 | 10 | 13 | 13 | 13
  CFB at Week 8, Follow-up | -1.20 (0.997) | -0.90 (0.953) | -0.38 (0.526) | -0.21 (1.218) | -0.34 (0.691)

3. Secondary Outcome: Number of Participants Who Achieved Hgb Response at Week 4
Description: Hgb response was defined as achieving an increase of at least 0.5 g/dL, 1.0 g/dL, 1.5 g/dL, and 2.0 g/dL in Hgb. The number of participants with Hgb response: Hgb increase <-1.0, Hgb increase -1.0 -< -0.5, Hgb increase -0.5 -< 0.5, Hgb increase 0.5 -< 1.0 and Hgb increase >=1.0 have been presented.
Time Frame: Week 4
Population: ITT population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 15 | 18 | 20 | 18 | 19
Participants
  Hgb increase <-1.0 | 11 | 4 | 3 | 0 | 0
  Hgb increase -1.0 -< -0.5 | 2 | 2 | 2 | 1 | 0
  Hgb increase -0.5 -< 0.5 | 2 | 10 | 8 | 7 | 6
  Hgb increase 0.5 -< 1.0 | 0 | 1 | 3 | 4 | 4
  Hgb increase >=1.0 | 0 | 1 | 4 | 6 | 9

4. Secondary Outcome: Percentage of Participants Who Achieved Hgb Response at Week 4
Description: Hgb response was defined as achieving an increase of at least 0.5 g/dL, 1.0 g/dL, 1.5 g/dL, and 2.0 g/dL in Hgb. The percentage of participants with Hgb response: Hgb increase <-1.0, Hgb increase -1.0 -< -0.5, Hgb increase -0.5 -< 0.5, Hgb increase 0.5 -< 1.0 and Hgb increase >=1.0 have been presented.
Time Frame: Week 4
Population: ITT population. Data for only those participants available at the indicated time points were collected and analyzed. Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 15 | 18 | 20 | 18 | 19
Percentage of participants
  Hgb increase <-1.0: number analyzed (Participants) | 15 | 18 | 20 | 0 | 0
  Hgb increase <-1.0 | 73 | 22 | 15 |  |
  Hgb increase -1.0 -< -0.5: number analyzed (Participants) | 15 | 18 | 20 | 18 | 0
  Hgb increase -1.0 -< -0.5 | 13 | 11 | 10 | 6 |
  Hgb increase -0.5 -< 0.5 | 13 | 56 | 40 | 39 | 32
  Hgb increase 0.5 -< 1.0: number analyzed (Participants) | 0 | 18 | 20 | 18 | 19
  Hgb increase 0.5 -< 1.0 |  | 6 | 15 | 22 | 21
  Hgb increase >=1.0: number analyzed (Participants) | 0 | 18 | 20 | 18 | 19
  Hgb increase >=1.0 |  | 6 | 20 | 33 | 47

5. Secondary Outcome: Number of Participants Who Reached Pre-defined Hgb Stopping Criteria
Description: Hgb stopping criteria was defined as: (1) Hgb <7.5 g/dL (2) 7.5 <= Hgb <1 3.0 g/dL and >2 g/dL Hgb change over 2W (3) Hgb >=13.0 g/dL. The number of participants who reached pre-defined Hgb stopping criteria have been presented.
Time Frame: Upto Week 4
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
Participants
  < 7.5 | 2 | 0 | 0 | 0 | 0
  7..5 -< 13.0 and >2 g/dL change | 0 | 0 | 0 | 2 | 1

6. Secondary Outcome: Maximum Observed CFB in Erythropoietin (EPO) Upto Week 4
Description: Blood samples for EPO were collected on Day 1 (pre-dose), Week 2 (collected approx 6-12 hours post-dose on arrival and after 1, 2 and 3 hours) and Week 4 (pre-dose and 3 hours post-dose). Maximum observed value meant maximum value between Week 1 and Week 4. Baseline was defined as the value on Day 1. Maximum observed CFB was calculated by subtracting the Baseline value from the maximum observed value between Week 1 and Week 4.
Time Frame: Baseline (Day 1) Upto Week 4
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units/liter
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 17 | 18 | 20 | 19 | 20
International units/liter | 6.658 (4.5414) | 34.951 (28.2718) | 94.518 (122.4985) | 151.012 (151.2964) | 173.446 (226.7241)

7. Secondary Outcome: Maximum Observed Percent CFB in Peak Vascular Endothelial Growth Factor (VEGF) Upto Week 4
Description: Blood samples for VEGF were collected on Day 1 (pre-dose), Week 2 (collected approximately 6-12 hours post-dose on arrival and after 1, 2 and 3 hours) and Week 4 (pre-dose and 3 hours post-dose). Maximum observed value meant maximum value between Week 1 and Week 4. Baseline was defined as the value on Day 1. Maximum observed percent CFB was calculated as 100 multiplied by the maximum observed exponential mean change on a log scale minus 1.
Time Frame: Baseline (Day 1) Upto Week 4
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 17 | 18 | 20 | 19 | 20
Percent change | 45.05 [1.00 to 108.32] | 18.78 [4.38 to 35.17] | 18.94 [8.19 to 30.75] | 27.70 [6.07 to 53.73] | 44.29 [14.44 to 81.94]

8. Secondary Outcome: Percent CFB in Hepcidine Upto Week 4
Description: Blood samples for hepcidine were collected on Day 1 (pre-dose), Week 2 (collected approximately 6-12 hours post-dose) and Week 4 (pre-dose). Baseline was defined as the value on Day 1. Percent CFB was calculated as 100 multiplied by the exponential mean change on a log scale minus 1.
Time Frame: Baseline (Day 1) Upto Week 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
Percent change
  Percent CFB in hepcidine,Week 2: number analyzed (Participants) | 17 | 18 | 20 | 19 | 20
  Percent CFB in hepcidine,Week 2 | 9.98 [-0.66 to 21.76] | -50.71 [-59.75 to -39.65] | -64.90 [-73.55 to -53.42] | -66.29 [-73.38 to -57.30] | -73.52 [-78.79 to -66.94]
  Percent CFB in hepcidine,Week 4: number analyzed (Participants) | 14 | 18 | 20 | 18 | 19
  Percent CFB in hepcidine,Week 4 | 3.26 [-9.18 to 17.42] | -60.34 [-67.40 to -51.76] | -69.66 [-77.38 to -59.30] | -69.06 [-77.57 to -57.31] | -77.71 [-82.08 to -72.28]

9. Secondary Outcome: CFB in Ferritin at Week 4
Description: Ferritin was used as marker of iron metabolism and utilization. Baseline was defined as the value on Day 1. CFB was calculated by subtracting the Baseline value from the post dose value at Week 4.
Time Frame: Baseline (Day 1) and Week 4
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms/liter
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 15 | 18 | 19 | 18 | 19
micrograms/liter | 4.7 (114.79) | -50.6 (40.28) | -78.3 (52.32) | -92.6 (107.07) | -113.3 (94.69)

10. Secondary Outcome: CFB in Total Iron Binding Capacity [TIBC], Unbound Iron Binding Capacity [UIBC] and Iron at Week 4
Description: TIBC, UIBC and Iron were used as marker of iron metabolism and utilization. Baseline was defined as the value on Day 1. CFB was calculated by subtracting the Baseline value from the post-dose value at Week 4.
Time Frame: Baseline (Day 1) and Week 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
micromoles/liter
  CFB in TIBC at Week 4: number analyzed (Participants) | 14 | 18 | 19 | 17 | 19
  CFB in TIBC at Week 4 | 0.2 (1.97) | 8.6 (3.96) | 14.4 (6.79) | 14.3 (5.67) | 17.2 (4.87)
  CFB in UIBC at Week 4: number analyzed (Participants) | 15 | 18 | 19 | 18 | 19
  CFB in UIBC at Week 4 | 0.8 (6.10) | 11.7 (6.61) | 19.2 (9.17) | 16.3 (9.18) | 22.1 (7.65)
  CFB in Iron at Week 4: number analyzed (Participants) | 15 | 18 | 19 | 18 | 19
  CFB in Iron at Week 4 | 0.0 (4.46) | -3.1 (4.96) | -4.8 (5.86) | -2.4 (7.16) | -4.9 (5.32)

11. Secondary Outcome: CFB in Transferrin at Week 4
Description: Transferrin was used as marker of iron metabolism and utilization. Baseline was defined as the value on Day 1. CFB was calculated by subtracting the Baseline value from the post-dose value at Week 4.
Time Frame: Baseline (Day 1) and Week 4
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 15 | 18 | 20 | 18 | 19
grams/liter | 0.041 (0.2013) | 0.449 (0.2958) | 0.626 (0.3605) | 0.677 (0.2948) | 0.804 (0.3944)

12. Secondary Outcome: Percent CFB in Transferrin Saturation (TS) at Week 4
Description: TS was used as marker of iron metabolism and utilization. Baseline was defined as the value on Day 1. Percent CFB was calculated as 100 multiplied by the exponential mean change on a log scale minus 1.
Time Frame: Baseline (Day 1) and Week 4
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 14 | 18 | 19 | 17 | 19
Percent change | 1.3 [-10.5 to 14.6] | -31.3 [-41.4 to -19.5] | -45.3 [-54.9 to -33.8] | -35.2 [-50.9 to -14.5] | -50.4 [-59.0 to -39.8]

13. Secondary Outcome: Plasma Pharmacokinetic Concentration of GSK1278863 and Metabolites (M) at Week 4
Description: Blood samples for plasma pharmacokinetic analysis were collected at Week 4 (pre-dose, 1, 2, 3 hours post-dose). Individual plasma GSK1278863 and M-GSK2391220, GSK2487818, GSK2506102, GSK2531398, GSK2531401, GSK2531403 concentrations have been presented.
Time Frame: Week 4
Population: Pharmacokinetic Population: All participants from whom a Pharmacokinetic sample was obtained and analyzed. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms/liter
Groups:
- GSK1278863 4 Milligrams (mg): Eligible participant's received GSK1278863 4 mg once daily for the 4 Week treatment period.
Arm/Group | Placebo | GSK1278863 4 Milligrams (mg) | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 0 | 19 | 20 | 19 | 20
micrograms/liter
  GSK1278863,Week 4,Pre-dose: number analyzed (Participants) | 0 | 18 | 19 | 18 | 18
  GSK1278863,Week 4,Pre-dose |  | 0.051 (NA) — Not estimated. | 0.031 (NA) — Not estimated. | 0.054 (NA) — Not estimated. | 0.767 (NA) — Not estimated.
  GSK1278863,Week 4,1 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK1278863,Week 4,1 hour Post-dose |  | 57.974 (86.6158) | 44.463 (64.5550) | 69.804 (104.4868) | 105.200 (109.5148)
  GSK1278863,Week 4,2 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK1278863,Week 4,2 hour Post-dose |  | 79.718 (68.6691) | 88.600 (97.6852) | 90.774 (95.5198) | 145.487 (148.5738)
  GSK1278863,Week 4,3 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK1278863,Week 4,3 hour Post-dose |  | 47.629 (38.0349) | 86.753 (73.4615) | 82.612 (91.3694) | 111.182 (104.4788)
  GSK2391220-M,Week 4,Pre-dose: number analyzed (Participants) | 0 | 18 | 19 | 18 | 18
  GSK2391220-M,Week 4,Pre-dose |  | 3.023 (2.4591) | 3.357 (1.8819) | 5.630 (6.2908) | 8.553 (8.1226)
  GSK2391220-M,Week 4,1 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2391220-M,Week 4,1 hour Post-dose |  | 2.105 (1.5209) | 2.883 (1.9924) | 4.340 (4.0699) | 8.417 (7.7174)
  GSK2391220-M,Week 4,2 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2391220-M,Week 4,2 hour Post-dose |  | 4.596 (3.2987) | 5.809 (4.6207) | 9.294 (7.6842) | 14.017 (10.5152)
  GSK2391220-M,Week 4,3 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2391220-M,Week 4,3 hour Post-dose |  | 6.444 (4.2038) | 8.227 (4.9024) | 11.116 (7.5314) | 17.216 (9.7376)
  GSK2487818-M,Week 4,Pre dose: number analyzed (Participants) | 0 | 18 | 19 | 18 | 18
  GSK2487818-M,Week 4,Pre dose |  | 0.141 (NA) — Not estimated. | 0.171 (0.1193) | 0.336 (0.6143) | 1.714 (5.1050)
  GSK2487818-M,Week 4,1 hour Post-dose: number analyzed (Participants) | 0 | 16 | 18 | 17 | 18
  GSK2487818-M,Week 4,1 hour Post-dose |  | 0.838 (1.0098) | 1.445 (1.9773) | 1.633 (2.4994) | 4.967 (6.2427)
  GSK2487818-M,Week 4,2 hour Post-dose: number analyzed (Participants) | 0 | 17 | 20 | 18 | 18
  GSK2487818-M,Week 4,2 hour Post-dose |  | 4.005 (3.2461) | 4.510 (4.4290) | 6.843 (6.4944) | 10.749 (8.8713)
  GSK2487818-M,Week 4,3 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 17
  GSK2487818-M,Week 4,3 hour Post-dose |  | 5.548 (3.7080) | 6.932 (4.5891) | 8.504 (5.9293) | 14.311 (7.8161)
  GSK2506102-M,Week 4,Pre-dose: number analyzed (Participants) | 0 | 18 | 19 | 18 | 18
  GSK2506102-M,Week 4,Pre-dose |  | 2.016 (0.7719) | 2.943 (1.0669) | 4.244 (2.8092) | 5.670 (2.2887)
  GSK2506102-M,Week 4,1 hour Post dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2506102-M,Week 4,1 hour Post dose |  | 1.159 (0.6277) | 1.705 (0.5636) | 2.473 (1.5656) | 3.552 (1.7551)
  GSK2506102-M,Week 4,2 hour Post dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2506102-M,Week 4,2 hour Post dose |  | 1.344 (0.6015) | 1.851 (0.8637) | 2.781 (1.6266) | 3.963 (2.0477)
  GSK2506102-M,Week4,3 hour Post dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2506102-M,Week4,3 hour Post dose |  | 1.569 (0.7467) | 2.163 (1.0410) | 3.045 (1.8790) | 4.382 (1.9892)
  GSK2531398-M,Week 4, Pre-dose: number analyzed (Participants) | 0 | 18 | 19 | 18 | 18
  GSK2531398-M,Week 4, Pre-dose |  | 0.717 (0.5356) | 0.772 (0.4409) | 1.478 (1.9681) | 2.496 (2.9738)
  GSK2531398-M,Week 4,1 hour Post-dos: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2531398-M,Week 4,1 hour Post-dos |  | 0.593 (0.4255) | 0.828 (0.6670) | 1.455 (1.7174) | 2.820 (2.8853)
  GSK2531398-M,Week 4,2 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2531398-M,Week 4,2 hour Post-dose |  | 1.715 (1.3986) | 2.141 (1.8332) | 3.496 (3.0818) | 5.318 (4.1121)
  GSK2531398-M,Week 4,3 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2531398-M,Week 4,3 hour Post-dose |  | 2.596 (1.5630) | 3.328 (2.1302) | 4.813 (3.4315) | 6.861 (3.7679)
  GSK2531401-M,Week 4, Pre-dose: number analyzed (Participants) | 0 | 18 | 19 | 18 | 18
  GSK2531401-M,Week 4, Pre-dose |  | 6.698 (3.9349) | 11.849 (6.4817) | 17.427 (11.3934) | 19.014 (7.8014)
  GSK2531401-M,Week 4,1 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2531401-M,Week 4,1 hour Post-dose |  | 3.426 (2.0445) | 6.383 (3.0760) | 9.259 (6.3198) | 11.288 (6.2673)
  GSK2531401-M,Week 4,2 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2531401-M,Week 4,2 hour Post-dose |  | 3.384 (1.6984) | 5.546 (2.7423) | 8.910 (5.2477) | 11.008 (6.8874)
  GSK2531401-M,Week 4,3 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2531401-M,Week 4,3 hour Post-dose |  | 3.911 (2.3475) | 5.849 (2.9144) | 8.864 (6.0433) | 11.417 (6.2311)
  GSK2531403-M,Week 4, Pre-dose: number analyzed (Participants) | 0 | 18 | 19 | 18 | 18
  GSK2531403-M,Week 4, Pre-dose |  | 5.609 (3.6494) | 8.183 (3.1169) | 12.703 (10.1144) | 16.524 (9.9794)
  GSK2531403-M,Week 4,1 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2531403-M,Week 4,1 hour Post-dose |  | 3.100 (2.0550) | 5.093 (1.9872) | 7.607 (5.5913) | 11.877 (8.2571)
  GSK2531403-M,Week 4,2 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2531403-M,Week 4,2 hour Post-dose |  | 4.857 (3.1705) | 6.906 (4.0374) | 10.755 (7.3841) | 15.573 (10.2857)
  GSK2531403-M,Week 4,3 hour Post-dose: number analyzed (Participants) | 0 | 18 | 20 | 18 | 18
  GSK2531403-M,Week 4,3 hour Post-dose |  | 6.320 (4.1558) | 8.744 (4.6123) | 12.119 (7.6702) | 18.369 (9.0090)

14. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE) on Therapy
Description: An AE is defined as any untoward medical occurrence in clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A SAE is defined as any AE which results in death; is life-threatening; requires participant hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event.
Time Frame: Upto Week 4
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 19 | 19 | 20 | 19 | 20
Participants
  Any AE | 5 | 6 | 8 | 7 | 5
  Any SAE | 1 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Chemistry and Hematology Data of Potential Clinical Importance (PCI) Upto Week 4
Description: The PCI range was as follows: alkaline phosphates >= 3 times upper limit of normal range [ULRR]), potassium (>0.5 millimoles/liter below the LLRR or >1.0 millimoles/liter above the ULRR), phosphate (>0.323 millimoles/liter above ULRR or below lower limit reference range [LLRR]), glucose (<3.9 or >22 millimoles/liter), magnesium (<LLRR or > 0.3 milimoles/liter above ULRR), lymphocytes <0.5x LLRR, neutrophils (<0.5 times LLRR), platelets (80 or >500 times giga/liter), platelets (80 or >500 times giga/liter) and leukocytes >1 x giga/liter below the LLRR or >5 x GI/L above the ULRR. The participants who had PCI values higher and lower than the reference range have been presented.
Time Frame: Upto Week 4
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 19 | 19 | 20 | 19 | 20
Participants
  Alkaline phosphatase, Week 4, High: number analyzed (Participants) | 18 | 18 | 19 | 18 | 19
  Alkaline phosphatase, Week 4, High | 0 | 1 | 0 | 0 | 0
  Potassium, High, Week 2: number analyzed (Participants) | 17 | 19 | 20 | 19 | 20
  Potassium, High, Week 2 | 0 | 0 | 0 | 1 | 0
  Potassium, High, Week 4: number analyzed (Participants) | 15 | 18 | 19 | 18 | 19
  Potassium, High, Week 4 | 1 | 0 | 0 | 1 | 0
  Phosphate, High, Week 2: number analyzed (Participants) | 17 | 19 | 20 | 19 | 20
  Phosphate, High, Week 2 | 1 | 9 | 10 | 7 | 9
  Phosphate, High, Week 4: number analyzed (Participants) | 18 | 18 | 19 | 18 | 19
  Phosphate, High, Week 4 | 2 | 9 | 11 | 8 | 10
  Potassium, low, Week 4: number analyzed (Participants) | 18 | 18 | 19 | 18 | 19
  Potassium, low, Week 4 | 0 | 0 | 1 | 0 | 0
  Potassium, low, Week 2: number analyzed (Participants) | 17 | 19 | 20 | 19 | 20
  Potassium, low, Week 2 | 0 | 0 | 1 | 0 | 0
  Glucose, Week 2, low: number analyzed (Participants) | 17 | 19 | 20 | 19 | 20
  Glucose, Week 2, low | 0 | 1 | 0 | 0 | 0
  Magnesium, low, Week 4: number analyzed (Participants) | 15 | 18 | 19 | 18 | 19
  Magnesium, low, Week 4 | 0 | 0 | 0 | 1 | 0
  Magnesium, low, Week 2: number analyzed (Participants) | 17 | 19 | 20 | 19 | 20
  Magnesium, low, Week 2 | 0 | 0 | 0 | 1 | 0
  Lymphocytes, low ,Week 1: number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
  Lymphocytes, low ,Week 1 | 0 | 0 | 0 | 1 | 0
  Lymphocytes, low ,Week 3: number analyzed (Participants) | 17 | 18 | 20 | 18 | 19
  Lymphocytes, low ,Week 3 | 0 | 0 | 1 | 0 | 0
  Neutrophils, low, Week 1: number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
  Neutrophils, low, Week 1 | 0 | 1 | 0 | 0 | 0
  Platelets, low, Week 1: number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
  Platelets, low, Week 1 | 0 | 0 | 1 | 0 | 0
  Platelets, low, Week 2: number analyzed (Participants) | 17 | 19 | 19 | 19 | 20
  Platelets, low, Week 2 | 0 | 0 | 1 | 0 | 0
  Platelets, low, Week 3: number analyzed (Participants) | 17 | 18 | 20 | 18 | 19
  Platelets, low, Week 3 | 0 | 0 | 1 | 0 | 0
  Platelets, low, Week 4: number analyzed (Participants) | 18 | 18 | 20 | 18 | 19
  Platelets, low, Week 4 | 0 | 0 | 1 | 0 | 0
  Leukocyte, low, Week 1: number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
  Leukocyte, low, Week 1 | 3 | 3 | 2 | 1 | 2
  Leukocyte, low, Week 2: number analyzed (Participants) | 17 | 19 | 19 | 19 | 20
  Leukocyte, low, Week 2 | 2 | 3 | 2 | 4 | 3
  Leukocyte, low, Week 3: number analyzed (Participants) | 17 | 18 | 20 | 18 | 19
  Leukocyte, low, Week 3 | 3 | 2 | 0 | 2 | 3
  Leukocyte, low, Week 4: number analyzed (Participants) | 18 | 18 | 20 | 18 | 19
  Leukocyte, low, Week 4 | 1 | 2 | 2 | 2 | 4

16. Secondary Outcome: Number of Participants With Vital Signs Parameters Systolic and Diastolic Blood Pressure (SBP,DBP) of PCI Upto Week 4
Description: Vital signs SBP and DBP were recorded pre-dialysis and post-dialysis. Measurements were taken from the participant while in a seated position or semi-supine in the dialysis chair. PCI range for SBP was < 85 or > 170 and for DBP was < 45 or > 100 millimeters of mercury. Participant's with values high and low from the PCI range have been presented.
Time Frame: Upto Week 4
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 19 | 19 | 20 | 19 | 20
Participants
  DBP, high, Pre-dialysis, Week 1: number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
  DBP, high, Pre-dialysis, Week 1 | 1 | 0 | 1 | 0 | 1
  DBP, high, Pre-dialysis, Week 2: number analyzed (Participants) | 17 | 19 | 20 | 19 | 20
  DBP, high, Pre-dialysis, Week 2 | 2 | 0 | 1 | 0 | 2
  DBP, high, Pre-dialysis,Week 4: number analyzed (Participants) | 18 | 18 | 20 | 18 | 19
  DBP, high, Pre-dialysis,Week 4 | 0 | 1 | 0 | 0 | 0
  DBP, high, Post-dialysis, Week 2: number analyzed (Participants) | 17 | 19 | 20 | 19 | 20
  DBP, high, Post-dialysis, Week 2 | 1 | 1 | 0 | 0 | 1
  DBP, high, Post-dialysis, Week 3: number analyzed (Participants) | 17 | 18 | 20 | 18 | 19
  DBP, high, Post-dialysis, Week 3 | 0 | 0 | 1 | 0 | 0
  DBP, high, Post-dialysis, Week 4: number analyzed (Participants) | 15 | 18 | 20 | 18 | 19
  DBP, high, Post-dialysis, Week 4 | 0 | 0 | 1 | 0 | 0
  DBP, low, Post-dialysis, Week 4: number analyzed (Participants) | 15 | 18 | 20 | 18 | 19
  DBP, low, Post-dialysis, Week 4 | 1 | 0 | 0 | 0 | 0
  SBP, high, Pre-dialysis, Week 1: number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
  SBP, high, Pre-dialysis, Week 1 | 2 | 4 | 0 | 3 | 1
  SBP, high, Pre-dialysis, Week 2: number analyzed (Participants) | 17 | 19 | 20 | 19 | 20
  SBP, high, Pre-dialysis, Week 2 | 4 | 3 | 3 | 2 | 4
  SBP, high, Pre dialysis, Week 3: number analyzed (Participants) | 17 | 18 | 20 | 18 | 19
  SBP, high, Pre dialysis, Week 3 | 2 | 3 | 2 | 2 | 1
  SBP, high, Pre-dialysis, Week 4: number analyzed (Participants) | 15 | 18 | 20 | 18 | 19
  SBP, high, Pre-dialysis, Week 4 | 2 | 6 | 1 | 4 | 2
  SBP, high, Post-dialysis, Week 1: number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
  SBP, high, Post-dialysis, Week 1 | 4 | 1 | 0 | 1 | 1
  SBP, high, Post-dialysis, Week 2: number analyzed (Participants) | 17 | 19 | 20 | 19 | 20
  SBP, high, Post-dialysis, Week 2 | 1 | 0 | 0 | 1 | 3
  SBP, high, Post-dialysis, Week 3: number analyzed (Participants) | 17 | 18 | 20 | 18 | 19
  SBP, high, Post-dialysis, Week 3 | 2 | 0 | 3 | 2 | 3
  SBP, high, Post-dialysis, Week 4: number analyzed (Participants) | 15 | 18 | 20 | 18 | 19
  SBP, high, Post-dialysis, Week 4 | 1 | 1 | 1 | 2 | 3
  SBP, low, Post-dialysis, Week 2: number analyzed (Participants) | 17 | 19 | 20 | 19 | 20
  SBP, low, Post-dialysis, Week 2 | 0 | 1 | 0 | 0 | 0
  SBP, low, Post-dialysis, Week 4: number analyzed (Participants) | 15 | 18 | 20 | 18 | 19
  SBP, low, Post-dialysis, Week 4 | 1 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Vital Sign Parameter Heart Rate (HR) of PCI Upto Week 4
Description: Vital sign HR was recorded pre-dialysis and post-dialysis. Measurements were taken from the participant while in a seated position or semi-supine in the dialysis chair. PCI range for HR was < 40 or > 110 beats per minute. Participant's with values higher than the PCI range have been presented.
Time Frame: Upto Week 4
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 19 | 19 | 20 | 19 | 20
Participants
  HR, high, Post-dialysis, Week 1: number analyzed (Participants) | 18 | 19 | 20 | 19 | 20
  HR, high, Post-dialysis, Week 1 | 0 | 0 | 1 | 0 | 0
  HR, high, Post-Dialysis, Week 3: number analyzed (Participants) | 17 | 18 | 20 | 18 | 19
  HR, high, Post-Dialysis, Week 3 | 0 | 0 | 1 | 0 | 0

18. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings Upto Week 4
Description: Full 12-lead ECGs included heart rate, PR, QRS, QT and QTc intervals. Measurements were taken from the participant while in a supine position. ECGs were performed consistently either before or after dialysis throughout the study. ECG abnormalities characterized as abnormal-not clinically significant (A-NCS) and abnormal-clinically significant (A-CS) upto W4 have been presented.
Time Frame: Upto Week 4
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
Number analyzed (Participants) | 19 | 19 | 20 | 19 | 20
Participants
  A-NCS, Week 2 | 5 | 8 | 6 | 7 | 7
  A-NCS, Week 4 | 2 | 8 | 5 | 8 | 6

ADVERSE EVENTS:
Time Frame: AEs were assessed from screening (Week 3-9) throughout the treatment period (4 Week) until follow-up (4 Weeks post the last dose of study medication).
Description: SAEs and nSAEs have been reported for the treatment period (4 Week). The safety population was used for analysis.
Groups:
- GSK1278863 4 mg: Eligible participant's received GSK1278863 4 mg once daily for the 4W treatment period.
- GSK1278863 6 mg: Eligible participant's received GSK1278863 6 mg once daily for the 4W treatment period.
- GSK1278863 8 mg: Eligible participant's received GSK1278863 8 mg once daily for the 4W treatment period.
- GSK1278863 10 mg: Eligible participant's received GSK1278863 10 mg once daily for the 4W treatment period.
Arm/Group | Placebo | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/20 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19 | 0/20 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 4/19 | 6/19 | 8/20 | 7/19 | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | GSK1278863 4 mg (N=19) | GSK1278863 6 mg (N=20) | GSK1278863 8 mg (N=19) | GSK1278863 10 mg (N=20)
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | GSK1278863 4 mg (N=19) | GSK1278863 6 mg (N=20) | GSK1278863 8 mg (N=19) | GSK1278863 10 mg (N=20)
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 2 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharyngitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Blister rupture (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Gastritis atrophic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.